CLINICAL TRIAL: NCT07068152
Title: COST-EFFECTIVENESS ANALYSIS OF "PIGGYBACK" TELENURSING IN THE IMMEDIATE PREOPERATIVE PERIOD OF ELECTIVE SURGERIES: RANDOMIZED CLINICAL TRIAL PROTOCOL
Brief Title: TELENURSING IN THE IMMEDIATE PREOPERATIVE PERIOD OF ELECTIVE SURGERIES
Acronym: TIPPES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Cintia Silva Fassarella, Advisor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TelenursingBR27
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Care; Telenursing; Patient Safety; Elective Surgical Procedures; Hospitals
Keywords: Elective Surgical Procedures; telenursing; patient safety; Preoperative Care; Hospitals
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Target of 176 patients for each arm of the research
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients in the intervention group will receive telenursing the day before surgery, with an immediate preoperative anamnesis script to be carried out by the main researcher. The following day, upon admission, before being transferred to the ward, the patient will be sent to the nursing assessment room, where the auxiliary researcher will apply the immediate preoperative anamnesis script in person.
  Interventions: Behavioral: Preoperative telenursing
- Control Group (No Intervention): Patients in the control group will not receive telenursing the day before surgery. Only the following day, upon admission, before being transferred to the ward, the patient will be sent to the nursing assessment room, where the auxiliary researcher will apply the immediate preoperative anamnesis script in person.

INTERVENTIONS:
Behavioral: Preoperative telenursing — The role of Nursing in Telenursing includes Nursing Consultation, Interconsultation, Consulting, Monitoring, Health Education and Reception of Spontaneous Demand mediated by Information and Communication Technologies. In this research, the researcher will make a telephone call the day before surgery to patients scheduled in the surgical map in order to guide them on immediate preoperative care.
  Other Names: Telehealth; eHealth; Telemedicine
  Arms: Intervention Group

SUMMARY:
Introduction: Telenursing encompasses Nursing Consultation, Interconsultation, Consulting, Monitoring, Health Education and Reception of Spontaneous Demand mediated by Information and Communication Technology. Objective: To perform a cost-effectiveness analysis of telenursing in the immediate preoperative period of adult patients undergoing elective surgeries in a university hospital of the SUS. Materials and method: Cost-effectiveness analysis nested in a clinical trial or empirical economic analysis of the piggyback evaluation type. Divided into 2 phases: a) Experimental research - randomized clinical trial to be carried out in a university hospital located in Rio de Janeiro and part of the SUS, with two parallel groups - intervention and control - with 1:1 allocation. The inclusion criteria will be adult patients, of both sexes, in the immediate preoperative period who are admitted on the day of elective surgery from their home. Patients who are hospitalized, patients in ophthalmology and obstetrics specialties, and those who will undergo examinations in the surgical center will be excluded. The sample size calculation was performed with a 95% confidence level and a sample loss of 5%, totaling 352 patients. The sampling will be random. Randomization and allocation concealment will be performed by the independent researcher. Patients in the GI will receive telenursing on the day before surgery with an anamnesis script for telenursing by the main researcher. On the day of surgery, all patients on the surgical map who came from their residence will be directed to the nursing assessment room where the auxiliary researcher will apply the in-person anamnesis script. The data will be processed by two independent researchers in an electronic spreadsheet and will be analyzed using descriptive and inferential statistics. The research will respect all legal and ethical frameworks necessary for its implementation; b) Prospective analysis of complete economic evaluation - in the piggyback evaluation modality - of the cost-effectiveness type. The effectiveness of telenursing will be verified by the outcome of surgical cancellation. A decision tree model will be used with a view to analyzing the SUS user at the local level (microcosting). The time horizon will be two days. The cost-effectiveness threshold will be 1 GDP per capita and the data analysis will include deterministic and probabilistic sensitivity. Expected results: It is expected to prove that telenursing can be a safe and efficient method for guiding patients before surgery, generating greater patient satisfaction, increasing access to information about health care for users through remote communication with nurses, reducing the waiting list by reducing surgical cancellations and possible incorporation of telenursing as a consolidated practice in the university hospital studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient recruitment will be conducted using the hospital's general surgical center surgical map. The participating population will consist of:
* All patients 18 years of age or older, of both sexes, in the immediate preoperative period;
* Admitted on the day of elective surgery;
* Coming from their home.

Exclusion Criteria:

* Inpatients;
* Ophthalmology, obstetrics, and pediatrics specialties;
* Exams performed in the surgical center, such as endoscopy, colonoscopy, video hysteroscopy, and others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Surgery cancellation | The researcher will verify it on the day after the surgery date
  The main outcome of this research is the surgery cancellation, which will be verified in the hospital's electronic system with its respective reason. This is a binary outcome.

SECONDARY OUTCOMES:
Inadequate immediate preoperative preparation | This will be verified at the time of the in-person nursing assessment on the day of surgery.
  Patients who fully comply with the instructions received the day before will be considered to have adequate surgical preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Cintia S Fassarella, Nurse, Principal Investigator — Postgraduate Program in Nursing at the State University of Rio de Janeiro
Locations (1):
- State University of Rio de Janeiro, Vila Isabel, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data that support the results of this research are anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication, no end date
Access Criteria: A proposal describing the planned analyses will be made available through publication in a data repository.

REFERENCES:
- [Background] Turunen E, Miettinen M, Setala L, Vehvilainen-Julkunen K. Elective Surgery Cancellations During the Time Between Scheduling and Operation. J Perianesth Nurs. 2019 Feb;34(1):97-107. doi: 10.1016/j.jopan.2017.09.014. Epub 2018 Apr 17. PMID 29678317
- [Background] McVey C. Telenursing: A Concept Analysis. Comput Inform Nurs. 2023 May 1;41(5):275-280. doi: 10.1097/CIN.0000000000000973. PMID 36223609
- [Background] Silva, L. de L. T., Souza, F. C. D. de, Coelho, K. R., & Araújo, S. S. Rate and causes of cancellation of elective surgeries in a hospital of Minas Gerais, Brazilian Journal of Development, 2021, 7, 77998-78011
- [Background] Silva Junior JM, Chaves RCF, Correa TD, Assuncao MSC, Katayama HT, Bosso FE, Amendola CP, Serpa Neto A, Malbouisson LMS, Oliveira NE, Veiga VC, Rojas SSO, Postalli NF, Alvarisa TK, Lucena BMN, Oliveira RAG, Sanches LC, Silva UVAE, Nassar Junior AP. Epidemiology and outcome of high-surgical-risk patients admitted to an intensive care unit in Brazil. Rev Bras Ter Intensiva. 2020 Mar;32(1):17-27. doi: 10.5935/0103-507x.20200005. Epub 2020 May 8. PMID 32401988
- [Background] Burguez Romero, L., Alves Ferreira, R., Bernardo Bueno, A. A., Duarte Pereira Silva Pinheiro, L., Silvestre Dos Santos Azevedo, A. P., Giron Camerini, F., De Mendonça Henrique, D., & Silva Fassarella, C., OUTPATIENT PREOPERATIVE TELECONSULTATION: NA INTEGRATIVE REVIEW, Revista Enfermagem Atual In Derme, 2023, 97, e023159
- [Background] Santos ML, Novaes CO, Iglesias AC. [Epidemiological profile of patients seen in the pre-anesthetic assessment clinic of a university hospital]. Rev Bras Anestesiol. 2017 Sep-Oct;67(5):457-467. doi: 10.1016/j.bjan.2016.06.002. Epub 2016 Aug 27. Portuguese. PMID 27576163
- [Background] Rocco M, Oliveira BL, Rizzardi DAA, Rodrigues G, Oliveira G, Guerreiro MG, Cruz VS, Naufel-Junior CR. Impact of the COVID-19 Pandemic on Elective and Emergency Surgical Procedures in a University Hospital. Rev Col Bras Cir. 2022 Aug 22;49:e20223324. doi: 10.1590/0100-6991e-20223324-en. eCollection 2022. PMID 36000684
- [Background] Pinheiro, Silvania Lopes; Vasconcelos, Raissa Ottes; Oliveira, João Lucas Campos de; Matos, Fabiana Gonçalves de Oliveira Azevedo; Tonini, Nelsi Salete; Alves, Débora Cristina Ignácio, Surgical cancellation rate: quality indicator at a public university hospital, REME rev. min. enferm, 2017, 21, e-1014.
- [Background] Pinheiro LDPS, Fassarella CS, Camerini FG, Henrique D de M, Ribeiro OMPL, Romero LB, Cancellation of outpatient surgery: an integrative review, Rev. enferm. UERJ, 2022, 30, 30:e66477
- [Background] Moura MSS, Carvalho SB, Braz ZR, Leal LB, Santos AMRD, Gouveia MTO, Avelino FVSD, Silva ARVD. Use of technologies by nurses to promote breastfeeding: a scoping review. Rev Esc Enferm USP. 2024 Feb 2;57:e20220466. doi: 10.1590/1980-220X-REEUSP-2022-0466en. eCollection 2024. PMID 38407608
- [Background] Lisboa LA, Mejia OAV, Arita ET, Guerreiro GP, Silveira LMVD, Brandao CMA, Dias RR, Dallan LRP, Miana L, Caneo LF, Jatene MB, Dallan LAO, Jatene FB. Impact of the First Wave of the COVID-19 Pandemic on Cardiovascular Surgery in Brazil: Analysis of a Tertiary Reference Center. Arq Bras Cardiol. 2022 Mar;118(3):663-666. doi: 10.36660/abc.20210235. No abstract available. English, Portuguese. PMID 35319617
- [Background] Islam, M. and Hossain, T. (2024) Exploring the Effects of Digital Transformation on Employees' Performance Management Systems of the Telecommunication Industry in Bangladesh. Journal of Human Resource and Sustainability Studies, 12, 289-314. doi: 10.4236/jhrss.2024.122016.
- [Background] Chua M, Lau XK, Ignacio J. Facilitators and barriers to implementation of telemedicine in nursing homes: A qualitative systematic review and meta-aggregation. Worldviews Evid Based Nurs. 2024 Jun;21(3):318-329. doi: 10.1111/wvn.12711. Epub 2024 Feb 10. PMID 38340069
- [Background] Bhanvadia RR, Carpinito GP, Kavoussi M, Lotan Y, Margulis V, Bagrodia A, Roehrborn CG, Gahan JC, Cadeddu J, Woldu S. Safety and Feasibility of Telehealth Only Preoperative Evaluation Before Minimally Invasive Robotic Urologic Surgery. J Endourol. 2022 Aug;36(8):1070-1076. doi: 10.1089/end.2021.0819. Epub 2022 Jul 5. PMID 35596562